# **COVER PAGE**

## **Document Type:**

Statistical Analysis Plan (SAP)

#### Official study title:

Computational Design, Fabrication, and Evaluation of Optimized Patient-Specific Transtibial Prosthetic Sockets

#### **NCT number:**

not yet assigned

#### **Document Date:**

02/15/2018

## Principal investigator:

Prof. Hugh Herr

## Sponsor:

NIH

## Participating sites:

Massachusetts Institute of Technology (MIT), Cambridge, MA, USA McGovern Institute for Brain Research, MIT, Cambridge, MA, USA

## Statistical analysis plan

Statistical analysis of the socket clinical evaluation data will focus on the following measurements:

- 1. local skin contact pressures
- 2. metabolic power
- 3. gait parameters (symmetry indices for joint angles, positions, torques, and ground reaction forces)
- 4. the socket evaluation questionnaire

For scalar comparisons a paired t-test, with the level of significance set at 0.05, will be used to test for differences between the novel and conventional sockets. For time-series analysis of variance (ANOVA) will be used.